CLINICAL TRIAL: NCT06094842
Title: A Phase I Safety and Feasibility Study of Cellular Immunotherapy for Extensive Stage Small Cell Neuroendocrine Prostate Cancer Using Autologous T Cells Lentivirally Transduced to Express L1CAM-Specific Chimeric Antigen Receptor
Brief Title: Autologous T Cells Lentivirally Transduced to Express L1CAM-Specific Chimeric Antigen Receptors in Treating Patients With Locally Advanced and Unresectable or Metastatic Small Cell Neuroendocrine Prostate Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study closed before opening to accrual
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1123589; NCI-2023-07464 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FH20229 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-10

CONDITIONS: Prostate Carcinoma; Prostate Small Cell Neuroendocrine Carcinoma; Stage III Prostate Cancer AJCC v8; Stage IV Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Bendamustine Hydrochloride; Biopsy; Specimen Handling; Bridge Therapy; Cyclophosphamide; fludarabine; Leukapheresis; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (autologous L1CAM-specific CAR+EGFRt+ T cells) (Experimental): Patients undergo leukapheresis to obtain PBMCs for T cell product manufacturing and may undergo bridging therapy at the discretion of the treating clinician on study. Patients then undergo lymphodepleting chemotherapy with cyclophosphamide IV and fludarabine IV on days -5, -4 and -33 or single agent bendamustine on days -4 and -3 at the discretion of the treating clinician and/or PI. Patients receive an autologous L1CAM-specific CAR+EGFRt+ T cells infusion on day 0. Based on disease response and persistence of CAR T cells, patients may receive additional lymphodepletion chemotherapy and an autologous L1CAM-specific CAR+EGFRt+ T cell infusion as soon as 6 weeks and no later than 24 weeks after the first infusion, or at the discretion of the PI. Patients also undergo ECHO or MUGA during screening. Patients undergo x-ray imaging, CT, bone scan, and blood sample collection throughout the trial. Additionally, patients may undergo tissue biopsy on the trial.
  Interventions: Drug: Bendamustine; Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Bridge Therapy; Procedure: Computed Tomography; Drug: Cyclophosphamide; Procedure: Echocardiography; Drug: Fludarabine; Procedure: Leukapheresis; Procedure: Multigated Acquisition Scan; Biological: T-cell Receptor-engineered T-cells; Procedure: X-Ray Imaging

INTERVENTIONS:
Drug: Bendamustine — Given IV
  Other Names: SDX-105
Procedure: Biopsy — Undergo tissue biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Bridge Therapy — Undergo bridging therapy
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B-518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719; WR-138719
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Biological: T-cell Receptor-engineered T-cells — Given autologous L1CAM-specific CAR+EGFRt+ T cells IV
  Other Names: T-cell Receptor-engineered T Cells; T-cell Receptor-engineered T-lymphocytes; TCR T Cells; TCR T-cells; TCR-engineered T-cells; TCR-modified T Cells
Procedure: X-Ray Imaging — Undergo chest x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase I trial studies the side effects and best dose of autologous CD8+ and CD4+ lentivirally transduced to express L1CAM-specific chimeric antigen receptor (CAR) and EGFRt mutation specific T cells and to see how well they work in treating patients with small cell neuroendocrine prostate cancer (SCNPC) that has spread to nearby tissue or lymph nodes (locally advanced) and cannot be removed by surgery (unresectable) or has spread from where it first started (primary site) to other places in the body (metastatic). CAR T-cell therapy is a type of treatment in which a patient's T cells (a type of immune system cell) are changed in the laboratory so they will attack tumor cells. T cells are taken from a patient's blood. Then the gene for a special receptor that binds to a certain protein on the patient's tumor cells is added to the T cells in the laboratory. Some solid tumor cells have an L1CAM protein on their surface, and T cells can be modified with a receptor, called a chimeric antigen receptor (CAR), to help recognize this protein and kill these tumor cells. Large numbers of the CAR T cells are grown in the laboratory and given to the patient by infusion for treatment of certain cancers. These L1CAM mutation specific T cells may help the body's immune system identify and kill L1CAM locally advanced and unresectable or metastatic small cell neuroendocrine prostate cancers' tumor cells.

DETAILED DESCRIPTION:
OUTLINE: This is a dose-escalation study of autologous L1CAM-specific CAR+EGFRt+ T cells.

Patients undergo leukapheresis to obtain peripheral blood mononuclear cells (PBMCs) for T cell product manufacturing and may undergo bridging therapy at the discretion of the treating clinician on study. Patients then undergo lymphodepleting chemotherapy with cyclophosphamide intravenously (IV) and fludarabine IV on days -5, -4 and -33 or single agent bendamustine on days -4 and -3 at the discretion of the treating clinician and/or principal investigator (PI). Patients receive an autologous L1CAM-specific CAR+EGFRt+ T cell infusion on day 0. Based on disease response and persistence of CAR T cells, patients may receive additional lymphodepletion chemotherapy and an autologous L1CAM-specific CAR+EGFRt+ T cell infusion as soon as 6 weeks and no later than 24 weeks after the first infusion, or at the discretion of the PI. Patients undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) during screening. Patients undergo x-ray imaging, computed tomography (CT), bone scan, and blood sample collection throughout the trial. Additionally, patients may undergo tissue biopsy on the trial.

After completion of study treatment, patients are followed up monthly for 3 months, then every 3 months up to 12 months then may undergo long-term follow-up annually for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥ 18 years of age
* Able to understand and give written informed consent
* Confirmation of small cell neuroendocrine prostate cancer (SCNPC) diagnosis by internal pathology review of initial or subsequent biopsy or other pathologic material at Fred Hutchinson Cancer Center/University of Washington
* Previously treated with a platinum-based chemotherapy regimen for SCNPC
* Participants may not have received prior therapy or plan to receive therapy (chemotherapy, immunotherapy and/or radiation therapy) or have undergone or plan to undergo major surgery within the last 3 weeks prior to leukapheresis AND initiation of lymphodepleting chemotherapy. Participants who have developed SCNPC in the context of prior androgen deprivation therapy (ADT) (i.e. medical/surgical castration) may continue on ADT at the discretion of their treating provider
* Evidence of L1CAM positivity by immunohistochemistry review of the patient's archival/fresh tumor samples
* Metastatic or locally advanced and unresectable disease
* Adequate performance status (Eastern Cooperative Oncology Group [ECOG] 0 or 1)
* Expected survival > 3 months
* Fertile participants must be willing to use an effective contraceptive method before, during, and for at least 4 months after the CAR T cell infusion
* Measurable disease per RECIST v1.1 criteria as determined by CT, MRI or positron emission tomography (PET) scan
* Hemoglobin > 9 g/dL (prior to leukapheresis)
* Absolute neutrophil count (ANC) > 1,500 per mm^3 (prior to leukapheresis)
* Platelets > 100,000 per mm^3 (prior to leukapheresis)
* Creatinine ≤ 1.5 x upper limit of normal (ULN) (prior to leukapheresis)
* Bilirubin ≤ 1.5 x ULN (≤ 3 x ULN in patients with known Gilbert's syndrome) (prior to leukapheresis)
* Aspartate transaminase (AST) ≤ 3.0 x ULN (prior to leukapheresis)
* Alanine transaminase (ALT) ≤ 3.0 x ULN (prior to leukapheresis)
* Alkaline phosphatase ≤ 3.0 x ULN (prior to leukapheresis)
* All prior treatment related toxicity prior to leukapheresis ≤ grade 2 by National Cancer Institute (NCI) Common Toxicity Criteria (CTC) version (v) 5.0

Exclusion Criteria:

* Participants with non-melanoma skin cancer are eligible, while participants with other prior malignancies must have had at least a 3-year disease-free interval
* Participants with active human immunodeficiency virus (HIV) (testing not required per protocol but status noted). Participants with adequately treated HIV will be permitted to enroll. Adequately treated HIV will be defined as being on a stable regimen of highly active anti-retroviral therapy (HAART), CD4 count ≥ 350 cells/mcL, undetectable viral load on standard polymerase chain reaction (PCR)-based testing and not requiring antibiotics or antifungal agents for the prevention of opportunistic infections
* Participants with active hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as HCV RNA is detected) infection. Participants with prior hepatitis B virus (HBV) infection are eligible. Participants with a history of hepatitis C virus (HCV) infection are eligible if they have been treated with curative intent and their hepatitis C PCR viral load is negative
* Known history of unstable angina or myocardial infarction (MI) within 6 months or clinically significant cardiac arrhythmia (other than stable atrial fibrillation) requiring anti-arrhythmia therapy
* New York Heart Association (NYHA) class III or IV congestive heart failure (CHF), clinically significant hypotension, uncontrolled symptomatic coronary artery disease, or a documented ejection fraction of < 35%
* Known history of clinically significant active chronic obstructive pulmonary disease (COPD), or other moderate-to-severe chronic respiratory illness present within 6 months
* Participants with clinically significant pulmonary dysfunction, as determined by medical history and physical exam should undergo pulmonary function testing. Those with an forced expiratory volume (FEV1) of < 50 % of predicted or diffusing capacity for carbon monoxide (DLCO) (corrected) < 40% will be excluded. Patients with > grade 1 dyspnea at rest or oxygen saturation < 94% on room air (resting)
* Infection requiring intravenous antibiotic use within 2 weeks of leukapheresis or uncontrolled active infection
* Baseline serum sodium level < 130 mEq/L
* Research participant is not receiving systemically administered steroid therapy. Physiologic glucocorticoid replacement therapy for management of adrenal insufficiency is allowed (≤ 10 mg daily of prednisone or equivalent)
* History of an autoimmune disease requiring immunosuppressant therapy within the past 5 years
* Other concurrent medical or psychiatric conditions that, in the investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations
* Known history of brain metastases.

  * Note: Brain imaging is not required to determine eligibility. However, this should be performed if there is clinical suspicion for brain metastases

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2028-03-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 12 months after last chimeric antigen receptor (CAR) T cell infusion
  The toxicities observed at each dose level will be summarized in terms of type (organ affected or laboratory determination such as absolute neutrophil count), severity (by National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version 5.0 and nadir or maximum values for the laboratory measures), date of onset and attribution. Tables will be created to summarize these toxicities and side effects by dose level.
Dose-limiting toxicity rates | Within 28 days of last CAR T cell infusion
  The toxicities observed at each dose level will be summarized in terms of type (organ affected or laboratory determination such as absolute neutrophil count), severity (by NCI CTCAE version 5.0 and nadir or maximum values for the laboratory measures), date of onset and attribution. Tables will be created to summarize these toxicities and side effects by dose level.

SECONDARY OUTCOMES:
Objective response | Up to 12 months after last CAR T cell infusion
  Will be determined using RECIST version 1.1 and will be summarized at each dose level, and the number and percent responding combined across dose levels.
Radiographic progression free survival | Up to 12 months after last CAR T cell infusion
  Will be assessed using RECIST v 1.1 criteria for soft tissue metastases and Prostate Cancer Working Group 3 criteria. Survival and time to relapse/progression will be summarized both by pooling across dose levels and within each dose level. Will calculate survival curves and the median expected survival duration, using the Kaplan-Meier estimate.
Overall survival | Up to 12 months after last CAR T cell infusion
  Will be assessed using RECIST v 1.1 criteria for soft tissue metastases and Prostate Cancer Working Group 3 criteria. Survival and time to relapse/progression will be summarized both by pooling across dose levels and within each dose level. Will calculate survival curves and the median expected survival duration, using the Kaplan-Meier estimate.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schweizer, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No